CLINICAL TRIAL: NCT00478192
Title: A Phase IIIb, Randomized, Double-Blind, Parallel Group, Multi-Center, Study to Assess the Efficacy and Safety of Multiple 30 Minute Infusions of YM087 (Conivaptan) in Subjects With Euvolemic or Hypervolemic Hyponatremia
Brief Title: Study of Efficacy & Safety for 3 Infusion Regimens of IV Conivaptan in Subjects With Euvolemic or Hypervolemic Hyponatremia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 087-CL-088
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Results first posted 2010-04-21 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-04

CONDITIONS: Hyponatremia
Keywords: hyponatremia; hypervolemic; euvolemic; edematous; conivaptan
MeSH Terms: conditions — Hyponatremia; Edema | interventions — conivaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regimen 1 Conivaptan QD (Experimental): 20 mg conivaptan once a day
  Interventions: Drug: Conivaptan
- Regimen 2 Conivaptan BID (Experimental): 20 mg conivaptan two times a day
  Interventions: Drug: Conivaptan
- Regimen 3 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Conivaptan — premix bag
  Other Names: YM087; Vaprisol
  Arms: Regimen 1 Conivaptan QD; Regimen 2 Conivaptan BID
Drug: Placebo — premix bag
  Arms: Regimen 3 Placebo

SUMMARY:
The study is designed to assess the efficacy and safety of multiple infusions of conivaptan in subjects with euvolemic or hypervolemic hyponatremia

ELIGIBILITY:
Inclusion Criteria:

* Euvolemic or hypervolemic (edematous) based on clinical presentation
* Serum sodium between 115 and 130mEq/L at baseline

Exclusion Criteria:

* Clinical presentation of volume depletion or dehydration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (23):
- United States (18):
  - Huntsville, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - Denver, Colorado
  - Jacksonville, Florida
  - Port Charlotte, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Hazard, Kentucky
  - Detroit, Michigan
  - Omaha, Nebraska
  - The Bronx, New York
  - Cincinnati, Ohio
  - Fairfield, Ohio
  - Toledo, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Orangeburg, South Carolina
- India (5):
  - Coimbatore
  - Indore
  - Jaipur
  - Karnāl
  - Visakhapatnam

REFERENCES:
- [Background] Koren MJ, Hamad A, Klasen S, Abeyratne A, McNutt BE, Kalra S. Efficacy and safety of 30-minute infusions of conivaptan in euvolemic and hypervolemic hyponatremia. Am J Health Syst Pharm. 2011 May 1;68(9):818-27. doi: 10.2146/ajhp100260. PMID 21515866
- See also: Link to Prescribing Information — http://www.astellas.us/docs/vaprisol.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient in the Placebo arm discontinued prior to dosing and therefore was not included in the Full Analysis Set (FAS) or the Safety Analysis Set (SAF).
Period: Overall Study
Arm/Group | Regimen 1 Conivaptan QD | Regimen 2 Conivaptan BID | Regimen 3 Placebo
Started | 20 | 20 | 10
Full Analysis Set / Safety Analysis Set | 20 | 20 | 9
End of Treatment | 18 | 16 | 8
Completed | 16 | 15 | 8
Not Completed | 4 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen 1 Conivaptan QD | Regimen 2 Conivaptan BID | Regimen 3 Placebo | Total
Number analyzed (Participants) | 20 | 20 | 9 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] — Population is Safety Analysis Set: All randomized patients who received at least one dose of study drug.
  years | 58.6 (17.36) | 67.5 (14.70) | 61.8 (20.19) | 62.8 (17.01)
Sex: Female, Male [Count of Participants; unit: Participants] — Population is Safety Analysis Set: All randomized patients who received at least one dose of study drug.
  Participants
    Female | 7 | 11 | 8 | 26
    Male | 13 | 9 | 1 | 23
Race/Ethnicity, Customized [Number; unit: participants] — Population is Safety Analysis Set: All randomized patients who received at least one dose of study drug.
  participants
    Asian | 7 | 4 | 3 | 14
    Black or African American | 1 | 1 | 2 | 4
    White | 12 | 15 | 4 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Sodium From Baseline to the 48 Hour Assessment or Study Drug Discontinuation.
Description: Baseline is the average of the two most recent serum sodium levels prior to start of dosing on day 1.
  Hour 48: Hour 48 or time that ended study participation prior to the hour 48 assessment.
  Change is calculated as Hour 48 - Baseline.
Time Frame: Baseline and 48 hours
Population: Full Analysis Set (FAS): all randomized patients who received at least one dose of study drug and who had baseline serum sodium data.
  The number of participants analyzed per arm represents FAS. The numbers of participants for each visit are noted in the category titles.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Regimen 1 Conivaptan QD | Regimen 2 Conivaptan BID | Regimen 3 Placebo
Number analyzed (Participants) | 20 | 20 | 9
mEq/L
  Baseline (N= 20; 20; 9) | 126.03 (4.017) | 126.39 (3.581) | 125.55 (3.648)
  Hour 48 (N=19; 17; 8) | 130.4 (5.21) | 133.4 (4.82) | 127.6 (2.36)
  Change from Baseline (N=19; 17; 8) | 4.00 (3.80) | 7.36 (4.04) | 1.16 (2.86)
Statistical Analysis 1: Comparison: Regimen 1 Conivaptan QD vs Regimen 2 Conivaptan BID; Statistical Analysis applies to "Change from Baseline"; Test type: Superiority or Other; p = 0.028, ANCOVA — P-Values are not adjusted on the basis of multiple comparrisons
Statistical Analysis 2: Comparison: Regimen 1 Conivaptan QD vs Regimen 3 Placebo; Statistical Analysis applies to "Change from Baseline"; Test type: Superiority or Other; p = 0.019, ANCOVA — P-Values are not adjusted on the basis of multiple comparrisons
Statistical Analysis 3: Comparison: Regimen 2 Conivaptan BID vs Regimen 3 Placebo; Statistical Analysis applies to "Change from Baseline"; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Values are not adjusted on the basis of multiple comparrisons

2. Secondary Outcome: Change From Baseline in Serum Sodium Level at Each Time Point Through the 48 Hour Assessment
Description: Baseline is the average of the two most recent serum sodium levels prior to start of dosing on day 1.
  Hour 48: Hour 48 or time that ended study participation prior to the hour 48 assessment.
  Change is calculated as Actual Data for each time point - Baseline
Time Frame: Baseline, Hour 4, Hour 12, Hour 16, Hour 24, Hour 28, Hour 36, Hour 40 and Hour 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Regimen 1 Conivaptan QD | Regimen 2 Conivaptan BID | Regimen 3 Placebo
Number analyzed (Participants) | 20 | 20 | 9
mEq/L
  Baseline (N=20; 20; 9) | 126.03 (4.02) | 126.39 (3.58) | 125.55 (3.65)
  Hour 4 (N=19; 20; 8) | 128.03 (4.62) | 128.47 (4.21) | 125.80 (4.63)
  Change at Hour 4 (N=19; 20; 8) | 1.59 (2.32) | 2.08 (2.65) | -0.63 (2.77)
  Hour 12 (N=19; 19; 7) | 128.22 (5.27) | 130.85 (5.88) | 127.21 (5.24)
  Change at Hour 12 (N=19; 19; 7) | 1.78 (3.44) | 4.65 (4.06) | 0.73 (3.92)
  Hour 16 (N=19; 17; 7) | 129.34 (4.51) | 131.04 (5.07) | 127.57 (3.78)
  Change at Hour 16 (N=19; 17; 7) | 2.90 (3.46) | 4.93 (3.28) | 1.09 (2.69)
  Hour 24 (N=18; 16; 8) | 128.87 (4.73) | 130.74 (5.33) | 127.48 (3.62)
  Change at Hour 24 (N=18; 16; 8) | 2.66 (3.76) | 4.62 (3.59) | 1.05 (2.73)
  Hour 28 (N=19; 17; 8) | 130.79 (4.94) | 131.62 (4.52) | 126.49 (4.03)
  Change at Hour 28 (N=19; 17; 8) | 4.35 (3.80) | 5.51 (2.75) | 0.06 (3.30)
  Hour 36 (N=19; 15; 8) | 131.42 (4.99) | 132.47 (5.04) | 127.31 (3.05)
  Change at Hour 36 (N=19; 15; 8) | 4.98 (3.73) | 6.54 (3.28) | 0.89 (2.55)
  Hour 40 (N=19; 16; 8) | 130.83 (5.04) | 132.23 (3.99) | 127.00 (1.85)
  Change at Hour 40 (N=19; 16; 8) | 4.39 (3.44) | 6.30 (3.27) | 0.58 (1.66)
  Hour 48 (N=19; 17; 8) | 130.44 (5.21) | 133.35 (4.82) | 127.59 (2.36)
  Change at Hour 48 (N=19; 17; 8) | 4.00 (3.80) | 7.36 (4.04) | 1.16 (2.86)

3. Secondary Outcome: Time From the First Dose of Study Medication to a Confirmed >4 mEq/L Increase From Baseline in Serum Sodium
Description: Confirmed sodium levels refers to two consecutive increases from baseline in sodium of >4 mEq/L; baseline is the average of the two most recent serum sodium levels prior to start of dosing on day 1.
  The endpoint was not evaluable in the placebo arm (median and interquartile range cannot be estimated) or the conivaptan QD arm (interquartile range cannot be estimated) because too high a percentage of patients were censored for the event. Only the conivaptan BID arm will be reported.
Time Frame: 48 Hours
Population: Full Analysis Set (FAS): all randomized patients who received at least one dose of study drug and who had baseline serum sodium data.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Regimen 2 Conivaptan BID
Number analyzed (Participants) | 20
Hours | 16.43 [12.00 to 32.00]

4. Secondary Outcome: Number of Patients With Confirmed Serum Sodium Level > 4 mEq/L Increase From Baseline Over 0 to 48 Hours
Description: Confirmed sodium levels refers to two consecutive increases from baseline in sodium of >4 mEq/L; baseline is the average of the two most recent serum sodium levels prior to start of dosing on day 1.
Time Frame: 48 Hours
Population: as for outcome 3
Measure: Number; unit: Patients
Arm/Group | Regimen 1 Conivaptan QD | Regimen 2 Conivaptan BID | Regimen 3 Placebo
Number analyzed (Participants) | 20 | 20 | 9
Patients | 12 | 17 | 2

5. Secondary Outcome: Number of Patients With Confirmed Serum Sodium Level Increase >6 mEq/L From Baseline or Confirmed Normal Serum Sodium Level (>135 mEq/L) Over the Duration 0 to 48 Hours
Description: Confirmed sodium levels refers to two consecutive increases from baseline in sodium of >6 mEq/L or two consecutive measurements >135 mEq/L; baseline is the average of the two most recent serum sodium levels prior to start of dosing on day 1.
Time Frame: 48 Hours
Population: as for outcome 3
Measure: Number; unit: Patients
Arm/Group | Regimen 1 Conivaptan QD | Regimen 2 Conivaptan BID | Regimen 3 Placebo
Number analyzed (Participants) | 20 | 20 | 9
Patients | 6 | 11 | 0

6. Secondary Outcome: Baseline -Adjusted Area Under the Curve (AUC) in Serum Sodium Over the Duration 0 to 48 Hours
Description: Each individual subject's change from baseline serum sodium levels was used to calculate baseline adjusted area under the curve serum sodium levels for a duration of Time 0 to Time t in hours (labeled as AUC(Na)(0-t). The last available serum sodium level prior to dosing on Day 1 was used as baseline.
  "t"=48 Hours
Time Frame: 48 Hours
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hour * mEq/L
Arm/Group | Regimen 1 Conivaptan QD | Regimen 2 Conivaptan BID | Regimen 3 Placebo
Number analyzed (Participants) | 20 | 20 | 9
Hour * mEq/L | 142.72 (132.94) | 244.17 (142.64) | 23.21 (91.49)
Statistical Analysis 1: Comparison: Regimen 1 Conivaptan QD vs Regimen 2 Conivaptan BID; Test type: Superiority or Other; p = 0.079, ANCOVA

7. Secondary Outcome: Change From Baseline in Effective Water Clearance (EWC) at Each Time Point Through the 48-hour Assessment
Description: Effective water clearence (EWC) was calculated as EWC=V(1-(Una+Uk)/(Pna+Pk)), where V is urine volume, Una is the urine sodium concentration, Uk is the urine potassium concentration, Pna is the serum/plasma sodium concentration, an Pk is the serum /plasma potassium concentration.
  Baseline is the average of the two most recent serum sodium levels prior to start of dosing on day 1.
  Hour 48: Hour 48 or time that ended study participation prior to the hour 48 assessment.
  Change is calculated as Actual Data for each time point - Baseline
Time Frame: Baseline, Hour 12, Hour 24,Hour 36 and Hour 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Regimen 1 Conivaptan QD | Regimen 2 Conivaptan BID | Regimen 3 Placebo
Number analyzed (Participants) | 20 | 20 | 9
mL
  Baseline (N=16; 12; 6) | 6.76 (47.91) | 39.86 (245.23) | 18.66 (45.05)
  Hour 12 (N=14; 12; 5) | 355.65 (684.35) | 405.21 (744.88) | 136.22 (154.94)
  Change at Hour 12 (N=12;12; 4) | 301.52 (671.78) | 365.35 (699.96) | 135.44 (123.36)
  Hour 24 (N=14; 12; 6) | -50.19 (794.22) | -261.27 (1009.24) | 368.01 (688.81)
  Change at Hour 24 (N=13; 11; 5) | -70.61 (796.01) | -391.76 (1206.39) | 383.73 (723.33)
  Hour 36 (N=15; 11; 6) | 36.85 (905.18) | 12.66 (743.24) | 726.96 (1013.78)
  Change at Hour 36 (N=12; 8; 5) | -91.07 (912.66) | -89.12 (805.36) | 810.45 (1079.89)
  Hour 48 (N=14; 11; 5) | -77.37 (1169.30) | -179.37 (852.58) | 569.09 (1392.07)
  Change at Hour 48 (N=12; 10; 4) | 80.23 (1116.99) | -240.39 (759.82) | 690.98 (2872.2)

8. Secondary Outcome: Change From Baseline in Free Water Clearance (FWC) at Each Time Point Through the 48-hour Assessment
Description: Free water clearance (FWC) was calculated as FWC=V(1-Uosm/Posm), where V is urine volume, Uosm is the urine osmolality, Posm is the plasma sodium osmolality.
  Baseline is the average of the two most recent serum sodium levels prior to start of dosing on day 1.
  Hour 48: Hour 48 or time that ended study participation prior to the hour 48 assessment.
  Change is calculated as Actual Data for each time point - Baseline
Time Frame: Baseline, Hour 24 and Hour 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Regimen 1 Conivaptan QD | Regimen 2 Conivaptan BID | Regimen 3 Placebo
Number analyzed (Participants) | 20 | 20 | 9
mL
  Baseline (N=14; 11; 6) | -53.87 (45.47) | 6.55 (165.07) | -34.90 (74.32)
  Hour 24 (N=14; 12; 6) | -972.29 (1455.66) | -611.14 (693.863) | -416.71 (666.97)
  Change at Hour 24 (N=11; 10; 5) | -936.99 (1618.46) | -513.33 (566.72) | -420.75 (747.84)
  Hour 48 (N=14;12; 5) | -1243.39 (2211.22) | -769.19 (934.31) | -592.96 (1050.94)
  Change at Hour 48 (N=11; 10; 4) | -1313.98 (2477.39) | -603.67 (761.90) | -702.11 (1117.92)

ADVERSE EVENTS:
Description: An Adverse Event was defined as treatment emergent if it occurred after the first dose of study drug through the ninth day after the last dose.
  Participants at Risk represent the Safety Analysis Set.
Arm/Group | Regimen 1 Conivaptan QD | Regimen 2 Conivaptan BID | Regimen 3 Placebo
Serious Adverse Events (participants affected / at risk) | 6/20 | 5/20 | 2/9
Other Adverse Events (participants affected / at risk) | 7/20 | 10/20 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 Conivaptan QD (N=20) | Regimen 2 Conivaptan BID (N=20) | Regimen 3 Placebo (N=9)
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Multi-organ failure (General disorders) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Coronary artery bypass (Surgical and medical procedures) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 Conivaptan QD (N=20) | Regimen 2 Conivaptan BID (N=20) | Regimen 3 Placebo (N=9)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1
Hypocoagulable state (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular arrthmia (Cardiac disorders) | 1 | 0 | 0
Hypothyrodism (Endocrine disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distention (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Bowel sounds abnormal (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Chest pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0
Hypothermia (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 2 | 0 | 0
Bronchitis chronic (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatine phosphokinaise increased (Investigations) | 0 | 0 | 1
Blood presure decreased (Investigations) | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0
Carotid bruit (Investigations) | 0 | 1 | 0
Chest X-ray abnormal (Investigations) | 1 | 0 | 0
Heart sounds abnormal (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 3 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the currency or completeness of the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.